CLINICAL TRIAL: NCT00511303
Title: Protein-Tyrosine Kinase Inhibitor (STI571) for Treatment of Patients With Ph+ Chronic Myeloid Leukemia Who Are Resistant to or Intolerant of *-Interferon. A Phase II Study
Brief Title: Protein-Tyrosine Kinase Inhibitor (STI571) for Treatment of Patients With Ph+ Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML 002
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2007-08-03 (Estimated); Status verified 2007-08

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Philadelphia chromosome; protein-tyrosine kinases
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: STI571

SUMMARY:
This is a Phase II, open-label, multi-center trial designed primarily to evaluate the rate of complete or major cytogenetic response of STI571 as demonstrated by a decrease in the percentage of Ph chromosome positive cells in the bone marrow, in patients with CML who are refractory to or intolerant of interferon-alpha.

During the core phase of the study, patients will receive once daily oral administration of STI571 at a dose of 400 mg, for up to 12 months. After completing 12 months of therapy patients may be eligible to receive additional therapy provided that, in the opinion of the investigator, the patient has benefited from treatment with STI571 and in the absence of safety concerns. Patients will receive STI571 on an outpatient basis.

During the extended phase (which is of indefinite duration), patients may continue STI571 until either progression to accelerated phase, blast phase, death, the development of intolerable toxicity, or the investigator feels it is no longer in the patient's best interest to continue therapy, whichever comes first. The number of visits will be at a reduced frequency. Patients who discontinue study drug will be followed for survival for up to 5 years.

STI571 will be considered active if the interferon-refractory patient population satisfies the target of achieving a complete or major response at a rate of at least 30%, within the preset error limits. Cytogenetic responses will be evaluated every three months and categorized as either complete (0% Ph+ chromosome cells), or major (1 to 35% Ph+ chromosome cells) responses. STI571 will be discontinued for any patient whose disease progresses to either the accelerated phase or blast crisis.

A minimum of 100 patients who are interferon refractory will receive STI571 administered at a dose of 400 mg once a day. In addition, the protocol is also open for patients who are intolerant to interferon-alpha in order to get a preliminary evaluation of their response to STI571 therapy. Up to 100 intolerant patients will be enrolled. Enrollment of intolerant patients will cease at 100, or whenever the 100 refractory patients are accrued, whichever comes first.

DETAILED DESCRIPTION:
This Phase II trial will evaluate at least 100 patients for the rate of complete or major cytogenetic response of STI571 as demonstrated by a decrease in the percentage of Ph chromosome positive cells in the bone marrow in patients with CML who are refractory to or intolerant of interferon-alpha. Statistical considerations are based on the refractory patient population only. Intolerant patients are included as long as recruitment of the refractory patients is ongoing, up to a maximum of 100 intolerant patients, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients * 18 years of age.
2. Patients with Ph chromosome positive CML in the chronic-phase of the disease.
3. Patients must have documented resistance to an interferon-alpha containing therapy, defined as any of the following:

   1. Hematologic Resistance - Failure to achieve a complete hematologic response, lasting for at least 1 month despite of 6 or more months of an interferon-alpha containing regimen.
   2. Cytogenetic Resistance - Bone marrow cytogenetics showing *65% Ph chromosome positivity after at least one year of interferon-alpha based therapy
   3. Cytogenetic Refractoriness - An increase in the Ph+ chromosome bone marrow cells by at least 30 percentage points (eg., from 20% to 50%, or from 30% to 60%) confirmed by two samples at least 1 month apart, or an increase to * 65%
   4. Hematologic Refractoriness - A rising WBC count (*100% increase and to a level *20 x 109/L confirmed by two samples taken at least two weeks apart) while receiving an interferon-alpha containing regimen.
4. Patients who have demonstrated intolerance to interferon-alpha therapy defined as: a documented * Grade 3 non-hematologic toxicity (grade 2 in case of neurologic or neuropsichiatric toxicity), persisting for more than 2 weeks, in a patient receiving an interferon-alpha containing regimen. Patients who are intolerant to interferon-alpha must be more than 3 months from time of diagnosis.
5. Written voluntary informed consent.

Exclusion Criteria:

1. Patients of childbearing potential without a negative pregnancy test prior to the initiation of study drug. Barrier contraceptive precautions are to be used throughout the trial in both sexes.
2. Serum bilirubin and creatinine concentrations more than twice the upper limit of the normal range.
3. SGOT and SGPT more than twice the upper limit of the normal range.
4. Percentage of blasts, or basophils in the peripheral blood or bone marrow > 15%.
5. Percentage of blasts plus promyelocytes in the peripheral blood or bone marrow ( 30%.
6. Patients with a platelet count < 100 x 109/L
7. Patients with an ECOG Performance Status Score * 3.
8. Patients receiving busulfan within 6 weeks of Visit 1.
9. Patients receiving treatment with interferon-alpha within 14 days of Visit 1.
10. Patients receiving treatment with cytosine arabinoside within 14 days of Visit 1.
11. Patients receiving treatment with hydroxyurea within 7 days of Visit 1.
12. Patients who have received other investigational agents within 28 days of Visit 1.
13. Patients with Grade 3/4 cardiac problems as defined by the New York Heart Association Criteria.
14. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable.
15. Patients who are likely to be submitted to any transplantation procedure during the study period (12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2000-08

PRIMARY OUTCOMES:
To determine the rate of complete and major cytogenetic response of STI571 as demonstrated by a decrease in the percentage of Ph chromosome positive cells in the bone marrow, in patients with CML who are refractory to interferon-alpha.

SECONDARY OUTCOMES:
To quantify the molecular response of STI571 as demonstrated by a decrease of bcr/abl transcript in peripheral blood cells,
To determine the rate and duration of complete hematological response,
To evaluate the duration of complete and major cytogenetic responses,
To evaluate the safety profile and improvement of symptomatic parameters,
To evaluate the time to accelerated disease, or blast crisis,
To evaluate overall survival,
To evaluate the rate and the duration of hematologic and cytogenetic response in patients intolerant to interferon-alpha

CONTACTS AND LOCATIONS:
Overall Officials: Michele Baccarani, MD, Principal Investigator — Istituto di Ematologia "L e A Seragnoli"-Policlinico S.Orsola-Malpighi di Bologna